CLINICAL TRIAL: NCT01792973
Title: HPV Infection and Cervical Lesions in HIV Infected Women in Thailand
Brief Title: HPV Infection and Cervical Lesions in HIV Infected Women in Thailand: A Prospective Study
Acronym: PapilloV
Status: Completed | Type: Observational
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: National Cancer Institute, France (Other Government); Fondation de France (Other)
Responsible Party: Principal Investigator, Marc Lallemant, Institut de Recherche pour le Developpement, Institut de Recherche pour le Developpement
Other Study IDs: PapilloV
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Cervical Cancer
Keywords: HIV; HPV; Women; Thailand; Antiretrovirals; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical secretions
Oversight: Data Monitoring Committee: Yes

SUMMARY:
HIV-infected women are at high risk of developing cervical cancer. This is a 3-year cohort study nested in the already existing Program for HIV Prevention and Treatment (PHPT) cohort of HIV-infected patients in Thailand (NCT 00433030). The main objective is to assess the prevalence, incidence, and clearance rate of HPV cervical infection and associated cervical lesion. The study will also provide the distribution of the HPV genotypes involved as well as other risk factors of cervical lesions. HIV-infected women receiving antiretrovirals, older than18 years of age, followed in the PHPT cohort or in the same hospitals are proposed to participate. An annual gynecological examination with a Pap-smear and a sampling for HPV testing is performed. Women with abnormal Pap-smear or with High-Risk HPV (HR-HPV) infection receive a more intensive follow-up with a colposcopy and a biopsy if necessary. Treatment is provided according to the National Guidelines.

DETAILED DESCRIPTION:
Title of the study: HPV Infection and Cervical Lesions in HIV infected Thai Women - A Prospective Study Country: Thailand Study period: 3 years Planned enrollment duration: 6 months

Primary objectives:

1. To evaluate the prevalence, the incidence, the persistence rate and the clearance rate of HPV cervical infection, of genotypes involved and of multiple infections.
2. To evaluate the prevalence, the incidence, the progression rate and the regression rate of cyto-histological abnormalities
3. To assess the efficacy of different screening algorithms using pap smear alone, pap-smear associated with HPV and HPV alone

Secondary objectives:

1. To determine the risk factors of high grade lesions (Cervical intraepithelial neoplasia (CIN)2 or higher) in HIV infected Thai women
2. To evaluate cyto-histology performances at different hospital levels Methods: A multicenter prospective cohort study nested in the PHPT cohort.

Inclusion criteria: HIV infected women, older than18 years of age, followed in the PHPT cohort or in the same hospitals.

Exclusion criteria: Virginity, total hysterectomy, pregnancy after 3rd month, inclusion in a HPV vaccination trial Planned number of patients to be enrolled: 884

Follow-up procedures:

Annual gynecological examination with a Pap-smear and a sampling for HPV testing is planned.

Women with abnormal Pap-smear or with High-Risk HPV (HR-HPV) infection will be referred to a colposcopist.

In case of abnormalities at the colposcopy, a biopsy will be performed.

* If the biopsy is normal or shows a CIN1, the women will be referred for a new colposcopic examination 6 months later.
* If the biopsy shows CIN2 or more, treatment will be provided -LEEP or conisation, or hysterectomy, and the women will be referred for a new colposcopic examination 6 months later.

Biological and pathological procedures:

* Pap-smears will be read by local pathologists in participating hospital.
* Biopsies will be read by local pathologists in participating hospital.
* HPV tests will all be performed in the PHPT virological laboratory in Chiang Mai.

Statistical methodology:

Descriptive statistics, univariate and multivariate analyses.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected women, older than 18 years of age, followed in the PHPT cohort

Exclusion Criteria:

* Virginity, total hysterectomy, pregnancy after 3rd month, inclusion in a HPV vaccination trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected women followed in the PHPT cohort
Sampling Method: Non-Probability Sample
Enrollment: 829 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
High risk HPV infection | January 2015
  HPV16, HPV18, HPV31, HPV33, HPV35, HPV39, HPV45, HPV51, HPV52, HPV56, HPV58, HPV59, HPV68
High grade cervical lesions | Up to 3 years
  Cervical intraepithelial neoplasia grade 2 or higher (CIN2+) in histology, and high grade squamous intraepithelial lesions or higher (HSIL+) in cytology

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Le Coeur, MD, PhD, Principal Investigator — Institut National d'Etudes Démographiques; Gonzague Jourdain, MD, PhD, Principal Investigator — Institut de Recherche pour le Developpement; Nicole Ngo-Giang- Huong, PharmaD, PhD, Principal Investigator — Institut de Recherche pour le Developpement; Isabelle Heard, MD, PhD, Principal Investigator — Centre national de réference des papillomavirus humains, Institut Pasteur; Aram Limtrakul, MD, Principal Investigator — Nakornping Hospital, Minsitry of Public Health; Nantasak Chotivanich, MD, Principal Investigator — Chonburi Hospital, Minsitry of Public Health; Chaiwat Putiyanun, MD, Principal Investigator — Chiang Kham Hospital, Ministry of Public Health; Samreung Rangdaeng, Associate professor, Principal Investigator — Department of Pathology Faculty of Medicine, Chiang Mai University
Locations (24):
- Thailand (24):
  - Prapokklao Hospital, Chanthaburi, Changwat Chanthaburi
  - Mae Chan Hospital, Mae Chan, Changwat Chiang Rai
  - Mae Sai Hospital, Mae Sai, Changwat Chiang Rai
  - Phan Hospital, Phan, Changwat Chiang Rai
  - Chonburi Hospital, Chon Buri, Changwat Chon Buri
  - Chiang Kham Hospital, Chiang Kham, Changwat Phayao
  - Buddhachinaraj Hospital, Phitsanulok, Changwat Phitsanulok
  - Hat Yai Hospital, Hat Yai, Changwat Songkhla
  - Lamphun Hospital, Lamphun, Chiang Mai
  - Nakornping Hospital, Mae Rim, Chiang Mai
  - Sanpatong Hospital, San Pa Tong, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai, Chiangrai
  - Mahasarakam Hospital, Maha Sarakham, Mahasarakam
  - Nakhonpathom Hospital, Nakhon Pathom, Nakhonpathom
  - Samutprakarn Hospital, Mueang Samut Prakan, Samutprakarn
  - Samutsakorn Hospital, Samut Sakhon, Samutsakorn
  - Bhumibol Adulyadej Hospital, Bangkok
  - Bhuddasothorn Hospital, Chachoengsao
  - Lampang Hospital, Lampang
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
  - Nong Khai Hospital, Nong Khai
  - Phayao Hospital, Phayao
  - Ratchaburi Hospital, Ratchaburi
  - Rayong Hospital, Rayong

REFERENCES:
- [Background] Dub T, Le Coeur S, Ngo-Giang-Huong N, Matanasarawut W, Suriyachai P, Saisawat K, Putiyanun C, Buranabanjasatean S, Leenasirimakul P, Randaeng S, Delory T. Prevalence of High-Risk Human Papillomavirus Infections before and after Cervical Lesion Treatment, among Women Living with HIV. J Clin Med. 2021 Jul 15;10(14):3133. doi: 10.3390/jcm10143133. PMID 34300302
- [Result] Le Coeur Sophie, Delory Tristan, Ngo-Giang-Huong Nicole, Rangdaeng Samreung, Heard Isabelle, Limtrakul Aram, Chotivanich Nantasak, Putiyanun Chaiwat, Leenasirimakul Prattana, Jourdain Gonzague. 2015. -"HPV Genotypes and factors associated with HR-HPV infection in HIV-infected women on Antiretroviral Therapy (ART) in Thailand: a national cohort". 30th International Papillomavirus Conference (HPV 2015), Lisbon, Portugal. 9-11 sept. 2015.
- [Result] Delory T, Ngo-Giang-Huong N, Rangdaeng S, Chotivanich N, Limtrakul A, Putiyanun C, Suriyachai P, Matanasarawut W, Jarupanich T, Liampongsabuddhi P, Heard I, Jourdain G, Lallemant M, Le Coeur S; PapilloV study group. Human Papillomavirus infection and cervical lesions in HIV infected women on antiretroviral treatment in Thailand. J Infect. 2017 May;74(5):501-511. doi: 10.1016/j.jinf.2017.02.007. Epub 2017 Feb 28. PMID 28254419